CLINICAL TRIAL: NCT00281632
Title: This Study is a Non-randomized, Open-label, Multi-center Phase II Study of GW786034 to Evaluate the Administration of Oral GW786034 in Subjects With Ovarian Cancer.
Brief Title: A Phase II, Open-Label Study Evaluating the Effect Of GW786034 In Subjects With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104450
Expanded Access: Available
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Results first posted 2011-01-04 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2011-02

CONDITIONS: Peritoneal Cancer; Ovarian Cancer; Neoplasms, Ovarian; Fallopian Tube Cancer
Keywords: Pazopanib; Fallopian tube cancer; Ovarian epithelial cancer; Peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — pazopanib

ARMS (1):
- Pazopanib (Experimental): 800 mg GW786034 administered orally on a daily basis.
  Interventions: Drug: GW786034

INTERVENTIONS:
Drug: GW786034 — 800 mg GW786034 administered orally on a daily basis.

SUMMARY:
This study was designed to find out how effective and safe GW786034, is in the treatment of epithelial ovarian, fallopian tube, or primary peritoneal cancer that has not responded to standard treatment.

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of epithelial ovarian, fallopian tube or primary peritoneal carcinoma.
* Has received one prior platinum-based chemotherapy regimen(cisplatin,carboplatin, or oxaliplatin).
* Has psychological, familial, sociological or geographical condition that does not permit compliance with the protocol.
* Is on a specifically prohibited medication or requires these medications during treatment with GW786034.

Exclusion criteria:

* Has had any surgery, chemotherapy, hormonal therapy, biologic, immunotherapy, or radiotherapy with in the last 28 days and has not recovered from such prior therapy.
* Poorly controlled hypertension(systolic 140mmHg or higher or Diastolic 90mmHg or higher).
* Currently taking warfarin.
* Low molecular weight heparin and low-dose warfarin(1mg per day)is permitted.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (9):
- United States (5):
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
- Australia (3):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Melbourne
- GSK Investigational Site, Singapore, Singapore

REFERENCES:
- [Background] Friedlander M, Hancock KC, Rischin D, Messing MJ, Stringer CA, Matthys GM, Ma B, Hodge JP, Lager JJ. A Phase II, open-label study evaluating pazopanib in patients with recurrent ovarian cancer. Gynecol Oncol. 2010 Oct;119(1):32-7. doi: 10.1016/j.ygyno.2010.05.033. Epub 2010 Jun 27. PMID 20584542

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib 800 mg: 800 milligrams (mg) pazopanib administered orally once daily
Period: Overall Study
Arm/Group | Pazopanib 800 mg
Started | 36
Completed | 0 (Three participants were ongoing in the study at the time of the data cut-off (30 Apr 2008).)
Not Completed | 36
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 2
Not completed — Disease Progression | 22
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Ongoing | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - South East Asian Heritage | 2
  White - White/Caucasian/European Heritage | 34

OUTCOME MEASURES:

1. Primary Outcome: Best Biochemical Response (Cancer Antigen [CA-125])
Description: Defined using modified Gynecologic Cancer Intergroup (GCIG) criteria: 50% response=≥50% decrease from baseline CA-125 (higher of 2 pretreatment CA-125 assessments) then confirmed after 21 days. 50% CA-125 response was normalized (CA-125 >21U/mL) or non-normalized (CA-125≤1U/mL). Progressive disease (PD) =CA-125 increase ≥100% from nadir (nadir >21U/mL) or ≥42U/mL (nadir ≤21U/mL); nadir was lowest CA-125. PD was confirmed after 21 days; otherwise=unconfirmed PD. Stable disease=scenarios that do not meet 50% response or PD. CA-125 response rate was defined as % of participants with 50% response.
Time Frame: Baseline to response (up to 3 years)
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 36
percentage of participants
  50% Response Normalized | 6
  50% Response Non-Normalized | 25
  Stable Disease | 56
  Progressive Disease | 3
  Unconfirmed Progressive Disease | 8
  Unknown | 3
Statistical Analysis 1: Comparison: Pazopanib 800 mg; Test type: Superiority or Other; Reponse rate = 31, 95% CI [16.3 to 48.1] — 50% Response Rate (Normalized and Non-Normalized)

2. Secondary Outcome: Time to Biochemical Response (CA-125)
Description: Time to biochemical response was calculated as the date pazopanib was first dosed to the date CA-125 was first reduced by 50% or greater. The reduction in CA-125 of 50% or greater was to be confirmed by a repeat measurement (no earlier than 21 days after initial evaluation documenting decrement). This was calculated for all participants with confirmed CA-125 50% reduction.
Time Frame: Baseline to response (up to 3 years)
Population: All participants with confirmed CA-125 50% reduction
Measure: Median (Full Range); unit: days
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 11
days | 29 [27 to 57]

3. Secondary Outcome: Duration of Biochemical Response (CA-125)
Description: Calculated as the date of confirmed first 50% or greater reduction in CA-125 to date of documented progression by clinical, radiographic, or biochemical criteria, whichever occurred earliest. This was calculated for all participants with confirmed CA-125 50% reduction.
Time Frame: Baseline to response (up to 3 years)
Population: All participants with confirmed CA-125 50% reduction
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 11
days | 113 [58.0 to 190.0]

4. Secondary Outcome: CA-125 Doubling Time Prior to and During Treatment With Pazopanib
Description: CA-125 doubling time is defined as the time for CA-125 to double from baseline value. This measure was not reported, as no participants had a post-baseline CA-125 that was double the baseline value. Therefore, the data did not warrant a report.
Time Frame: Baseline to doubling of CA-125 (up to 3 years)
Population: All participants with confirmed CA-125 50% reduction
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Response and Stable Disease (SD)
Description: Overall response and stable disease (SD) are based on biochemical, radiographic, and clinical assessments according to the modified criteria of Gynecologic Cancer Intergroup (GCIG) (see primary outcome). Response is presented as the percentage of participants with the given response.
Time Frame: Baseline to response (up to 3 years)
Population: All participants
Measure: Number; unit: percentage of participants
Groups:
- Pazopanib 800 mg With Measurable Disease: Participants with measureable disease at baseline who were administered 800 milligrams (mg) pazopanib administered orally once daily
- Pazopanib 800 mg Without Measurable Disease: Participants without measureable disease at baseline who were administered 800 milligrams (mg) pazopanib administered orally once daily.
- Pazopanib 800 mg All: All participants administered 800 milligrams (mg) pazopanib administered orally once daily
Arm/Group | Pazopanib 800 mg With Measurable Disease | Pazopanib 800 mg Without Measurable Disease | Pazopanib 800 mg All
Number analyzed (Participants) | 17 | 19 | 36
percentage of participants
  Complete Reponse | 0 | 5.3 | 2.8
  Partial Response | 17.6 | 15.8 | 16.7
  Stable Disease | 17.6 | 26.3 | 22.2
  Progressive Disease | 64.7 | 47.4 | 55.6
  Unknown | 0 | 5.3 | 2.8
Statistical Analysis 1: Comparison: Pazopanib 800 mg With Measurable Disease; Test type: Superiority or Other; Response rate = 17.6, 95% CI [3.8 to 43.4] — Response rate (CR+PR)
Statistical Analysis 2: Comparison: Pazopanib 800 mg Without Measurable Disease; Test type: Superiority or Other; Response rate = 21.1, 95% CI [6.1 to 45.6] — Response rate (CR+PR)
Statistical Analysis 3: Comparison: Pazopanib 800 mg All; Test type: Superiority or Other; Response rate = 19.4, 95% CI [8.2 to 36.0] — Response rate (CR+PR)

6. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Progression-free survival analysis was performed on all participants and then stratified by CA-125 response status (having confirmed 50% reduction or not). PFS was defined as the time from the date of the first dose of study drug to the date of documented and confirmed progression by clinical, radiographic, or biochemical criteria, whichever occurred earliest, or to date of death due to any causes.
Time Frame: Date of the first dose of study drug to the date of documented and confirmed progression by clinical, radiographic, or biochemical criteria, whichever occurred earliest, or to date of death due to any causes (up to 2 years)
Population: All participants with PFS
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Pazopanib 800 mg Responders: 800 milligrams (mg) pazopanib administered orally once daily Responders
- Pazopanib 800 mg Non-Responders: 800 milligrams (mg) pazopanib administered orally once daily Non-Responders
- Pazopanib 800 mg All: 800 milligrams (mg) pazopanib administered orally once daily All participants
Arm/Group | Pazopanib 800 mg Responders | Pazopanib 800 mg Non-Responders | Pazopanib 800 mg All
Number analyzed (Participants) | 10 | 20 | 30
days | 168 [84.0 to 217.0] | 57 [51.0 to 85.0] | 84 [57.0 to 141.0]

7. Secondary Outcome: Overall Tumor Response
Description: Overall tumor response following daily administration of pazopanib was defined using radiographic assessments based on Response Evaluation Criteria for Solid Tumors (RECIST) criteria for subjects with measurable disease at baseline.
Time Frame: Baseline to response (up to 3 years)
Population: All participants
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 17
participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 5
  Progressive Disease | 10
  Unknown | 2

8. Secondary Outcome: Number of Participants With the Indicated Maximum Shift From Baseline (BL) in Diastolic Blood Pressure
Description: Summary of shifts in diastolic blood pressure from baseline to the maximum change in the study. mmHg, millimeters of mercury.
Time Frame: Baseline to response (up to 3 years)
Population: All participants. Data are presented for only those participants who provided measurements at baseline and maximum shift post-baseline.
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 36
participants
  BL, 50-89 mmHg; shift to post-BL, <50 mmHg | 0
  BL, 50-89 mmHg; shift to post-BL, 50-89 mmHg | 16
  BL, 50-89 mmHg; shift to post-BL, 90-109 mmHg | 16
  BL, 50-89 mmHg; shift to post-BL, >=109 mmHg | 0
  BL, 90-109 mmHg; shift to post-BL, <50 mmHg | 0
  BL, 90-109 mmHg; shift to post-BL, 50-89 mmHg | 3
  BL, 90-109 mmHg; shift to post-BL, 90-109 mmHg | 1
  BL, 90-109 mmHg; shift to post-BL, >=109 mmHg | 0

9. Secondary Outcome: Number of Participants With the Indicated Maximum Shift From Baseline (BL) in Systolic Blood Pressure
Description: Summary of shifts in systolic blood pressure from baseline to the maximum change in the study. mmHg, millimeters of mercury.
Time Frame: Baseline to response (up to 3 years)
Population: as for outcome 8
Measure: Number; unit: participants
Groups:
- Pazopanib 800 mg: : 800 milligrams (mg) pazopanib administered orally once daily
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 36
participants
  BL, 90-139 mmHg; shift to post-BL, <90 mmHg | 0
  BL, 90-139 mmHg; shift to post-BL, 90-139 mmHg | 13
  BL, 90-139 mmHg; shift to post-BL, 140-169 mmHg | 16
  BL, 90-139 mmHg; shift to post-BL, >=170 mmHg | 2
  BL, 140-169 mmHg; shift to post-BL, <90 mmHg | 0
  BL, 140-169 mmHg; shift to post-BL, 90-139 mmHg | 0
  BL, 140-169 mmHg; shift to post-BL, 140-169 mmHg | 5
  BL, 140-169 mmHg; shift to post-BL, >=170 mmHg | 0
  BL, >=170 mmHg; shift to post-BL, 90-139 mmHg | 0
  BL, >=170 mmHg; shift to post-BL, 140-169 mmHg | 0
  BL, >=170 mmHg; shift to post-BL, >=170 mmHg | 0

10. Secondary Outcome: Number of Participants With the Indicated Maximum Shift From Baseline (BL) in Heart Rate
Description: Summary of shifts in heart rate from baseline to the maximum change in the study. bpm, beats per minute.
Time Frame: Baseline to response (up to 3 years)
Population: All participants
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 36
participants
  BL, 44-100 bpm; shift to post-BL, <44 bpm | 0
  BL, 44-100 bpm; shift to post-BL, 44-100 bpm | 32
  BL, 44-100 bpm; shift to post-BL, 101-120 bpm | 3
  BL, 44-100 bpm; shift to post-BL, >120 bpm | 0
  BL, 101-120 bpm; shift to post-BL, <44 bpm | 0
  BL, 101-120 bpm; shift to post-BL, 44-100 bpm | 1
  BL, 101-120 bpm; shift to post-BL, 101-120 bpm | 0
  BL, 101-120 bpm; shift to post-BL, >120 bpm | 0

11. Secondary Outcome: Mean Change From Baseline to Response in Albumin
Description: Change from baseline is calculated as the value at the time of response minus the value at Baseline.
Time Frame: Baseline to response (up to 3 years)
Population: All participants. Data are presented for only those participants who provided chemistry measurements at both baseline and the time of response.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 29
grams per liter (g/L) | -1.5 (8.82)

12. Secondary Outcome: Mean Change From Baseline to Response in Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, and Lactate Dehydrogenase
Description: Change from baseline is calculated as the value at the time of response minus the value at Baseline.
Time Frame: Baseline to response (up to 3 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: International Units per liter (IU/L)
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 29
International Units per liter (IU/L)
  Alkaline phosphatase, n=29 | 7.3 (27.76)
  Alanine aminotransferase, n=29 | 13.0 (23.25)
  Aspartate aminotransferase, n=28 | 7.1 (12.65)
  Lactate dehydrogenase, n=21 | 4.62 (29.630)

13. Secondary Outcome: Mean Change From Baseline to Response in Amylase and Lipase
Description: Change from baseline is calculated as the value at the time of response minus the value at Baseline.
Time Frame: Baseline to response (up to 3 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 22
Units per liter (U/L)
  Amylase | 7.32 (31.038)
  Lipase | 7.273 (24.994)

14. Secondary Outcome: Mean Change From Baseline to Response in Total Bilirubin and Creatinine
Description: Change from baseline is calculated as the value at the time of response minus the value at Baseline.
Time Frame: Baseline to response (up to 3 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micromoles per liter (umol/l)
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 29
micromoles per liter (umol/l)
  Total bilirubin | 0.715 (2.7039)
  Creatinine | 1.37 (8.846)

15. Secondary Outcome: Mean Change From Baseline to Response in Calcium, Glucose, Potassium, Sodium, and Urea
Description: Change from baseline is calculated as the value at the time of response minus the value at Baseline.
Time Frame: Baseline to response (up to 3 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/l)
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 29
millimoles per liter (mmol/l)
  Calcium, n=29 | -0.038 (0.1034)
  Glucose, n=28 | 0.302 (1.7285)
  Potassium, n=28 | -0.02 (0.553)
  Sodium, n=29 | 0.1 (2.85)
  Urea, n=29 | -0.227 (1.3410)

16. Secondary Outcome: Mean Change From Baseline to Response in Thyroxine
Description: Change from baseline is calculated as the value at the time of response minus the value at Baseline.
Time Frame: Baseline to response (up to 3 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/l)
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 2
nanomoles per liter (nmol/l) | 0.003 (0.0018)

17. Secondary Outcome: Mean Change From Baseline to Response in Thyroid Stimulating Hormone
Description: Change from baseline is calculated as the value at the time of response minus the value at Baseline.
Time Frame: Baseline to response (up to 3 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milliunits per liter (MU/L)
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 24
milliunits per liter (MU/L) | 0.87 (1.693)

18. Secondary Outcome: Mean Change From Baseline to Response in Hemoglobin and Hematocrit
Description: Change from baseline is calculated as the value at the time of response minus the value at Baseline.
Time Frame: Baseline to response (up to 3 years)
Population: All participants. Data are presented for only those participants who provided hematology measurements at both baseline and the time of response.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 30
g/L
  Hemoglobin | -0.53 (13.952)
  Hematocrit | -0.00 (0.048)

19. Secondary Outcome: Mean Change From Baseline to Response in Lymphocytes, Neutrophils, Platelet Count, and White Blood Count
Description: Change from baseline is calculated as the value at the time of response minus the value at Baseline.
Time Frame: Baseline to response (up to 3 years)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: giga (10^9) per liter (GI/L)
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 30
giga (10^9) per liter (GI/L)
  Lymphocytes | 0.32 (2.191)
  Neutrophils | -0.12 (2.276)
  Platelet count | -9.93 (75.487)
  White blood cell count | -0.28 (2.373)

ADVERSE EVENTS:
Arm/Group | Pazopanib 800 mg
Serious Adverse Events (participants affected / at risk) | 6/36
Other Adverse Events (participants affected / at risk) | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=36)
Constipation (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Hepatic enzyme increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Breast cancer situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary retention (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=36)
Diarrhea (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 5
Abdominal distensions (Gastrointestinal disorders) | 4
Ascites (Gastrointestinal disorders) | 4
Abdominal pain lower (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 17
Edema peripheral (General disorders) | 3
Malaise (General disorders) | 2
Mucosal inflammation (General disorders) | 2
Pain (General disorders) | 2
Pyrexia (General disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Alanine aminotransferase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 9
Gamma-glutamyltransferase increased (Investigations) | 6
Blood alkaline phosphastase (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
Headache (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hair color changes (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 11
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Anemia (Blood and lymphatic system disorders) | 2
Lymph node pain (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Insomnia (Psychiatric disorders) | 4
Tinnitus (Ear and labyrinth disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.